CLINICAL TRIAL: NCT00784719
Title: A Phase I/II Prospective, Randomized, Double Masked, Vehicle And Comparator Controlled, Dose Ranging Study Of CP-690,550 In Subjects With Dry Eye Disease.
Brief Title: A Prospective, Randomized, Placebo and Active Comparator Controlled Study of CP-690,550 in Subjects With Dry Eye.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921034; A3921034
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — tofacitinib; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment 1 (Experimental)
  Interventions: Drug: CP-690,550
- Treatment 2 (Experimental)
  Interventions: Drug: CP-690,550
- Treatment 3 (Experimental)
  Interventions: Drug: CP-690,550
- Treatment 4 (Experimental)
  Interventions: Drug: CP-690,550
- Active comparator (Active Comparator)
  Interventions: Drug: Cyclosporine
- Placebo (Placebo Comparator)
  Interventions: Drug: CP-690,550 Vehicle

INTERVENTIONS:
Drug: CP-690,550 — Ophthalmic topical solution, low dose, dosed at least once/day, 8 weeks
  Arms: Treatment 1
Drug: CP-690,550 — Ophthalmic topical solution, medium dose, dosed at least once/day, 8 weeks
  Arms: Treatment 2
Drug: CP-690,550 — Ophthalmic topical solution, intermediate dose, dosed at least once/day, 8 weeks
  Arms: Treatment 3
Drug: CP-690,550 — Ophthalmic topical solution, high dose, dosed at least once/day, 8 weeks
  Arms: Treatment 4
Drug: Cyclosporine — Ophthalmic topical solution, 0.05%, dosed at least once/day, 8 weeks
  Arms: Active comparator
Drug: CP-690,550 Vehicle — Ophthalmic topical solution, dosed at least once/day, 8 weeks
  Arms: Placebo

SUMMARY:
A prospective, randomized, placebo and active comparator controlled study of CP-690,550 in subjects with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of dry eye for at least 6 months.
* Signs of moderate to severe dry eye

Exclusion Criteria:

* Women who are nursing or pregnant
* Participation in other studies within 30 days of screening visit
* Ocular disorders that may confound interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (25):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Artesia, California
  - Pfizer Investigational Site, Centennial, Colorado
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Morrow, Georgia
  - Pfizer Investigational Site, Roswell, Georgia
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lynbrook, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, High Point, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Liew MS, Zhang M, Kim E, Akpek EK. Prevalence and predictors of Sjogren's syndrome in a prospective cohort of patients with aqueous-deficient dry eye. Br J Ophthalmol. 2012 Dec;96(12):1498-503. doi: 10.1136/bjophthalmol-2012-301767. Epub 2012 Sep 21. PMID 23001257
- [Derived] Huang JF, Yafawi R, Zhang M, McDowell M, Rittenhouse KD, Sace F, Liew SH, Cooper SR, Pickering EH. Immunomodulatory effect of the topical ophthalmic Janus kinase inhibitor tofacitinib (CP-690,550) in patients with dry eye disease. Ophthalmology. 2012 Jul;119(7):e43-50. doi: 10.1016/j.ophtha.2012.03.017. Epub 2012 May 18. PMID 22607938
- [Derived] Liew SH, Nichols KK, Klamerus KJ, Li JZ, Zhang M, Foulks GN. Tofacitinib (CP-690,550), a Janus kinase inhibitor for dry eye disease: results from a phase 1/2 trial. Ophthalmology. 2012 Jul;119(7):1328-35. doi: 10.1016/j.ophtha.2012.01.028. Epub 2012 Apr 22. PMID 22525048
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921034&StudyName=A%20prospective%2C%20randomized%2C%20placebo%20and%20active%20comparator%20controlled%20study%20of%20CP-690%2C550%20in%20subjects%20with%20dry%20eye.%20%20%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Twice Daily: One drop (45 microliter [mcL]) of matching placebo solution twice daily in each eye for 8 weeks.
- CP-690,550, 0.0003% Twice Daily: One drop (45 mcL) of 0.0003 percent (%) CP-690,550 solution twice daily in each eye for 8 weeks.
- CP-690,550, 0.001% Twice Daily: One drop (45 mcL) of 0.001% CP-690,550 solution twice daily in each eye for 8 weeks.
- CP-690,550, 0.003% Twice Daily: One drop (45 mcL) of 0.003% CP-690,550 solution twice daily in each eye for 8 weeks.
- CP-690,550, 0.005% Twice Daily: One drop (45 mcL) of 0.005% CP-690,550 solution twice daily in each eye for 8 weeks.
- CP-690,550, 0.005% Once Daily: One drop (45 mcL) of 0.005% CP-690,550 solution once daily in the morning in each eye and 1 drop of matching placebo once daily in the evening in each eye for 8 weeks.
- Restasis Twice Daily: One drop (45 mcL) of Restasis (cyclosporine) 0.05% ophthalmic emulsion twice daily in each eye for 8 weeks.
Period: Overall Study
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Started | 47 | 46 | 47 | 48 | 48 | 44 | 47
Completed | 44 | 43 | 46 | 48 | 42 | 41 | 42
Not Completed | 3 | 3 | 1 | 0 | 6 | 3 | 5
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 2 | 1 | 1 | 0 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily | Total
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47 | 327
Age Continuous [Mean (Standard Deviation); unit: years] | 62.3 (12.54) | 59.5 (11.57) | 60.7 (11.73) | 58.7 (14.57) | 59.9 (11.69) | 59.8 (14.83) | 58.9 (14.25) | 60.0 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 40 | 34 | 39 | 37 | 38 | 255
  Male | 15 | 11 | 7 | 14 | 9 | 7 | 9 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Systemic Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Systemic AEs are the events which are not localized but occur throughout the systemic circulation.
Time Frame: Baseline up to Week 8
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
percentage of participants | 27.7 | 8.7 | 29.8 | 27.1 | 18.8 | 18.2 | 23.4

2. Primary Outcome: Percentage of Participants With Ocular Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Ocular AEs are the events which are localized in the ocular region.
Time Frame: Baseline up to Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
percentage of participants | 25.5 | 21.7 | 31.9 | 22.9 | 22.9 | 22.7 | 36.2

3. Primary Outcome: Percentage of Participants With Ocular Tolerability Assessment
Description: Ocular tolerability assessment included evaluation of severity and duration of the 5 symptoms: burning/stinging, blurred vision, ocular discomfort, pain, tearing. Severity was assessed on a 4-point scale, where 0=none, 1=mild, 2=moderate and 3=severe. Duration was assessed as immediate (if subsided within 5 minutes [<5 min] after application) or persistent (if continued beyond 5 minutes [>=5 min] after application).
Time Frame: Baseline up to Week 8
Population: ITT population included all enrolled participants who received at least one dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 46 | 47 | 48 | 47 | 43 | 44
percentage of participants
  Ocular discomfort:none | 55.6 | 50.0 | 53.2 | 52.1 | 46.8 | 69.8 | 34.1
  Ocular discomfort:mild | 33.3 | 28.3 | 25.5 | 29.2 | 44.7 | 18.6 | 34.1
  Ocular discomfort:moderate | 11.1 | 19.6 | 19.1 | 14.6 | 8.5 | 9.3 | 25.0
  Ocular discomfort:severe | 0.0 | 2.2 | 2.1 | 4.2 | 0.0 | 2.3 | 6.8
  Ocular discomfort:moderate/severe, duration>=5 min | 4.4 | 10.9 | 8.5 | 10.4 | 4.3 | 7.0 | 22.7
  Burning sensation:none | 26.7 | 43.5 | 23.4 | 33.3 | 29.8 | 32.6 | 18.2
  Burning sensation:mild | 55.6 | 39.1 | 59.6 | 39.6 | 53.2 | 48.8 | 40.9
  Burning sensation:moderate | 17.8 | 15.2 | 14.9 | 22.9 | 14.9 | 16.3 | 36.4
  Burning sensation:severe | 0.0 | 2.2 | 2.1 | 4.2 | 2.1 | 2.3 | 4.5
  Burning sensation:moderate/severe,duration>=5 min | 0.0 | 2.2 | 2.1 | 0.0 | 4.3 | 4.7 | 11.4
  Pain:none | 82.2 | 80.4 | 80.9 | 85.4 | 85.1 | 88.4 | 61.4
  Pain:mild | 13.3 | 10.9 | 8.5 | 6.3 | 12.8 | 7.0 | 25.0
  Pain:moderate | 4.4 | 6.5 | 6.4 | 6.3 | 2.1 | 2.3 | 9.1
  Pain:severe | 0.0 | 2.2 | 4.3 | 2.1 | 0.0 | 2.3 | 4.5
  Pain:moderate/severe, duration >=5 min | 2.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Tearing:none | 55.6 | 63.0 | 68.1 | 72.9 | 66.0 | 69.8 | 47.7
  Tearing:mild | 40.0 | 26.1 | 21.3 | 16.7 | 29.8 | 11.6 | 29.5
  Tearing:moderate | 4.4 | 10.9 | 10.6 | 10.4 | 4.3 | 18.6 | 11.4
  Tearing:severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 11.4
  Tearing:moderate/severe, duration >= 5 min | 0.0 | 2.2 | 6.4 | 2.1 | 0.0 | 4.7 | 6.8
  Blurred vision:none | 51.1 | 54.3 | 53.2 | 58.3 | 51.1 | 44.2 | 36.4
  Blurred vision:mild | 40.0 | 30.4 | 34.0 | 27.1 | 36.2 | 34.9 | 40.9
  Blurred vision:moderate | 6.7 | 15.2 | 12.8 | 8.3 | 8.5 | 18.6 | 20.5
  Blurred vision:severe | 2.0 | 0.0 | 0.0 | 6.3 | 4.3 | 2.3 | 2.3
  Blurred vision:moderate/severe, duration >=5 min | 0.0 | 2.2 | 4.3 | 4.2 | 6.4 | 7.0 | 2.3

4. Primary Outcome: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 10 Millimeter (mm) Schirmer Wetting Score Without Anesthesia at Week 8
Description: Schirmer test without anesthesia: well standardized test used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac for 5 min. The length of wetting was recorded to the nearest 0.5 millimeter (mm). If the wetting line was oblique, halfway point was used. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. Last observation carried forward (LOCF) was the method used for imputing missing data at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 45 | 47 | 48 | 46 | 44 | 45
percentage of participants | 20.0 | 17.8 | 25.5 | 18.8 | 26.1 | 27.3 | 35.6

5. Secondary Outcome: Time to Achieve >= 10mm Schirmer Test Score Without Anesthesia
Description: Schirmer test without anesthesia: well standardized test used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac for 5 min. The length of wetting was recorded to the nearest 0.5 mm. If the wetting line was oblique, halfway point was used. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline through Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
days | NA [NA to NA] — Median and corresponding upper limit of 80% confidence interval (CI) were not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding upper limit of 80% CI were not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis. | 59.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 58.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | NA [NA to NA] — Median and corresponding upper limit of 80% CI were not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis. | 57.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | NA [NA to NA] — Median and corresponding upper limit of 80% CI were not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis.
Statistical Analysis 1: Comparison: CP-690,550, 0.001% Twice Daily; Test type: Superiority or Other; Median = 59.00, 80% CI 2-sided [lower limit 57.0] (Upper limit of 80% CI was not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis.)
Statistical Analysis 2: Comparison: CP-690,550, 0.003% Twice Daily; Test type: Superiority or Other; Median = 58.00, 80% CI 2-sided [lower limit 58.0] (Upper limit of 80% CI was not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis.)
Statistical Analysis 3: Comparison: CP-690,550, 0.005% Once Daily; Test type: Superiority or Other; Median = 57.00, 80% CI 2-sided [lower limit 29.0] (Upper limit of 80% CI was not estimable as there were insufficient number of participants, who achieved >=10 mm Schirmer test score in this reporting group, for the analysis.)

6. Secondary Outcome: Time to Achieve 100 Percent (%) Clearance of Corneal Staining
Description: Corneal staining was assessed by instilling sodium fluorescein dye in the eye and after 1 to 2 minutes, observing for corneal staining with the aid of a yellow filter and slit lamp. The cornea was divided into five different zones and each corneal zone was graded independently using a 0 to 3 grading scale; where 0=none, 1=slight, 2=moderate, 3=severe. Results from study eye were to be reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline through Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
days | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis. | NA [NA to NA] — Median and corresponding 80% CI were not estimable as there were insufficient number of participants, who achieved 100% clearance of corneal staining in this reporting group, for the analysis.

7. Secondary Outcome: Time to Achieve >= 5 Units Decrease in Ocular Comfort Index (OCI) Score
Description: OCI: validated questionnaire to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contained 12 questions, each measured on a 7-point Likert scale ranging from 0 (never) to 6 (always/severe). Total score was transformed to range of 0 to 100, higher score indicated more ocular discomfort. Negative change from baseline indicated improvement.
Time Frame: Baseline through Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
days | 15.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 8.50 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 15.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 9.50 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 9.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 15.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study. | 16.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated as it was corresponding to type I error of 10% (1-sided) specified for the study.
Statistical Analysis 1: Comparison: Placebo Twice Daily; Test type: Superiority or Other; Median = 15.00, 80% CI 2-sided [9.0 to 28.0]
Statistical Analysis 2: Comparison: CP-690,550, 0.0003% Twice Daily; Test type: Superiority or Other; Median = 8.50, 80% CI 2-sided [8.0 to 27.0]
Statistical Analysis 3: Comparison: CP-690,550, 0.001% Twice Daily; Test type: Superiority or Other; Median = 15.00, 80% CI 2-sided [15.0 to 27.0]
Statistical Analysis 4: Comparison: CP-690,550, 0.003% Twice Daily; Test type: Superiority or Other; Median = 9.50, 80% CI 2-sided [8.0 to 15.0]
Statistical Analysis 5: Comparison: CP-690,550, 0.005% Twice Daily; Test type: Superiority or Other; Median = 9.00, 80% CI 2-sided [8.0 to 15.0]
Statistical Analysis 6: Comparison: CP-690,550, 0.005% Once Daily; Test type: Superiority or Other; Median = 15.00, 80% CI 2-sided [8.0 to 43.0]
Statistical Analysis 7: Comparison: Restasis Twice Daily; Test type: Superiority or Other; Median = 16.00, 80% CI 2-sided [15.0 to 30.0]

8. Secondary Outcome: Change From Baseline in Schirmer Wetting Score Without Anesthesia at Week 1, 2, 4, 6 and 8
Description: as for outcome 5
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. LOCF method was used for imputing missing data at Week 8. Here, 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
mm
  Baseline (n=47,46,47,48,48,44,47) | 4.15 (2.07) | 4.40 (2.20) | 4.02 (2.12) | 3.77 (1.87) | 4.43 (2.29) | 4.40 (2.24) | 4.74 (2.03)
  Change at Week 1 (n=45,45,47,47,44,42,43) | 2.06 (4.54) | 1.68 (4.69) | 0.80 (3.03) | 2.07 (3.87) | 1.80 (4.64) | 2.68 (6.11) | 3.60 (5.44)
  Change at Week 2 (n=44,46,46,48,45,44,44) | 2.43 (4.98) | 1.63 (4.04) | 2.67 (4.44) | 3.13 (4.61) | 2.74 (4.60) | 3.43 (6.62) | 3.84 (5.66)
  Change at Week 4 (n=44,43,45,48,44,39,43) | 2.42 (6.64) | 2.69 (4.56) | 2.56 (4.76) | 1.72 (3.60) | 1.66 (5.03) | 4.21 (7.03) | 4.06 (6.65)
  Change at Week 6 (n=43,44,43,47,42,41,43) | 1.86 (3.82) | 1.41 (3.27) | 1.59 (3.55) | 1.76 (4.11) | 3.64 (6.57) | 4.65 (6.30) | 3.87 (5.75)
  Change at Week 8 (n=45,46,47,48,47,44,45) | 1.89 (5.22) | 2.30 (4.73) | 2.19 (4.22) | 3.59 (6.22) | 2.60 (4.80) | 3.76 (6.28) | 4.48 (7.05)

9. Secondary Outcome: Change From Baseline in Schirmer Wetting Score With Anesthesia at Week 8
Description: Schirmer test was performed 2 to 3 minutes after 1 drop of proparacaine 0.5% was placed in lower conjunctival fornix and superior bulbar conjunctiva of each eye. It was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac for 5 min. The length of wetting was recorded to the nearest 0.5 mm. If the wetting line was oblique, halfway point was used. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline, Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 43 | 47
mm
  Baseline (n=47,46,47,48,48,43,47) | 6.56 (4.69) | 7.58 (4.44) | 6.63 (5.05) | 6.67 (4.01) | 7.85 (5.35) | 7.92 (5.13) | 8.14 (5.75)
  Change at Week 8 (n=43,43,45,48,41,39,42) | 2.24 (5.07) | 0.13 (5.47) | 2.56 (6.11) | 1.48 (5.48) | -0.44 (5.13) | 0.83 (6.04) | 1.74 (5.74)

10. Secondary Outcome: Percentage of Participants Who Achieved >=10 mm Schirmer Wetting Score Without Anesthesia at Week 1, 2, 4 and 6
Description: as for outcome 5
Time Frame: Week 1, 2, 4, 6
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) included those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 45 | 47 | 48 | 44 | 44 | 44
percentage of participants
  Week 1 | 20.0 | 9.1 | 6.4 | 14.9 | 11.6 | 16.7 | 30.2
  Week 2 | 18.2 | 20.0 | 23.9 | 16.7 | 25.0 | 22.7 | 36.4
  Week 4 | 18.2 | 20.9 | 17.8 | 10.4 | 16.3 | 28.2 | 30.2
  Week 6 | 20.9 | 9.1 | 16.3 | 12.8 | 34.1 | 39.0 | 34.9

11. Secondary Outcome: Percentage of Participants Who Achieved >=10 mm Schirmer Wetting Score With Anesthesia at Week 8
Description: as for outcome 9
Time Frame: Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 43 | 43 | 45 | 48 | 41 | 39 | 42
percentage of participants | 32.6 | 27.9 | 48.9 | 31.3 | 24.4 | 25.6 | 38.1

12. Secondary Outcome: Change From Baseline in Corneal Staining Scores at Week 1, 2, 4, 6 and 8
Description: Corneal staining was assessed using fluorescein dye, a yellow filter, and a slit lamp. The cornea was divided into 5 different zones. Each corneal zone was graded independently using a 0 to 3 grading scale; where 0=none, 1=slight, 2=moderate, 3=severe. Sum of scores of each zone led to total score. Total score range: 0 to 15, higher score indicated greater staining. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
units on a scale
  Baseline (n=47,46,47,48,48,44,47) | 6.64 (3.45) | 5.63 (1.95) | 5.83 (2.10) | 6.73 (2.94) | 6.21 (2.54) | 6.36 (2.71) | 6.85 (3.50)
  Change at Week 1 (n=45,45,47,47,44,42,44) | -1.16 (2.39) | -0.89 (2.05) | -0.87 (2.25) | -1.32 (2.58) | -0.20 (1.95) | -1.17 (2.51) | 0.02 (3.27)
  Change at Week 2 (n=44,46,46,48,45,44,44) | -1.02 (3.16) | -1.15 (2.33) | -1.00 (2.19) | -1.98 (2.50) | -0.91 (2.26) | -1.52 (2.73) | -0.61 (2.94)
  Change at Week 4 (n=44,43,45,48,44,39,43) | -2.48 (2.53) | -1.02 (2.58) | -1.33 (2.69) | -1.40 (2.54) | -0.82 (2.45) | -2.10 (2.31) | -1.00 (2.86)
  Change at Week 6 (n=43,44,43,48,42,41,43) | -2.21 (3.49) | -1.39 (2.50) | -1.21 (2.42) | -1.75 (3.06) | -1.31 (3.00) | -2.27 (2.69) | -1.49 (3.03)
  Change at Week 8 (n=45,46,47,48,47,44,45) | -2.67 (3.44) | -1.39 (2.92) | -1.28 (2.65) | -1.58 (3.04) | -1.47 (2.73) | -2.64 (2.94) | -1.18 (3.50)

13. Secondary Outcome: Percentage of Participants Who Demonstrated 100% Clearance of Corneal Staining
Description: Corneal staining was assessed using fluorescein dye, yellow filter, slit lamp. Cornea was divided into 5 different zones. Each corneal zone was graded independently using 0 to 3 grading scale:0=none, 1=slight, 2=moderate, 3=severe. Sum of scores of each zone led to total score. Total score range: 0 to 15, higher score indicated greater staining. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Week 1, 2, 4, 6, 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. LOCF method was used for imputing missing data at Week 8. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 46 | 47 | 48 | 48 | 44 | 44
percentage of participants
  Week 1 | 2.2 | 0.0 | 0.0 | 0.0 | 0.0 | 4.8 | 0.0
  Week 2 | 2.3 | 4.3 | 0.0 | 4.2 | 0.0 | 4.5 | 0.0
  Week 4 | 4.5 | 2.3 | 4.4 | 6.3 | 2.3 | 2.6 | 4.7
  Week 6 | 4.7 | 6.8 | 7.0 | 4.2 | 7.1 | 7.3 | 7.0
  Week 8 | 6.7 | 6.5 | 4.3 | 10.4 | 6.4 | 15.9 | 4.5

14. Secondary Outcome: Change From Baseline in Interpalpebral Conjunctival Staining Score at Week 1, 2, 4, 6 and 8
Description: Interpalpebral conjunctival staining was performed 1 minute following ocular administration of lissamine green dye with aid of slit lamp. Based on Oxford grading system, bulbar conjunctiva was divided into 2 zones: nasal, temporal. Staining were graded using a 6-point scale (0=absent, 5=severe). Total score=sum of 2 zone scores. Total score range: 0 to 10, higher score=higher damage to eyes due to dryness. Negative change from baseline indicated improvement. Results from study eye are reported. Study eye is the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: ITT population. LOCF method was used for imputing missing data at Week 8. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 43 | 47
units on a scale
  Baseline (n=47,46,47,48,48,43,47) | 2.77 (2.36) | 2.17 (1.43) | 2.21 (1.81) | 2.38 (2.08) | 2.17 (1.99) | 1.91 (1.66) | 2.43 (2.03)
  Change at Week 1 (n=45,45,47,47,44,42,43) | -0.44 (1.52) | -0.38 (1.76) | -0.34 (1.75) | -0.13 (2.06) | -0.45 (1.42) | 0.17 (1.50) | -0.09 (1.92)
  Change at Week 2 (n=44,46,46,48,45,43,44) | -0.89 (1.53) | -0.26 (1.41) | -0.37 (1.44) | -0.29 (1.57) | -0.44 (1.62) | -0.19 (1.38) | 0.05 (2.47)
  Change at Week 4 (n=44,43,45,48,44,39,43) | -1.11 (1.86) | -0.53 (1.65) | -0.60 (1.56) | -0.27 (1.87) | -0.11 (1.37) | 0.18 (1.35) | -0.07 (1.64)
  Change at Week 6 (n=43,44,43,48,42,41,43) | -0.84 (1.38) | -0.73 (1.63) | -0.44 (1.74) | -0.46 (1.68) | -0.12 (1.71) | 0.02 (1.98) | -0.14 (1.90)
  Change at Week 8 (n=45,46,47,48,47,43,45) | -0.82 (2.01) | -0.57 (1.78) | -0.62 (1.81) | -0.63 (1.71) | -0.13 (1.78) | -0.14 (1.82) | -0.18 (1.57)

15. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT) at Week 1, 2, 4, 6 and 8
Description: TBUT was the time interval between the last complete blink and the first appearance of a dry spot, or disruption in the tear film. It was measured under a slit lamp following instillation of fluorescein dye in the eye using a stopwatch. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. LOCF method was used for imputing missing data at Week 8. 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
seconds
  Baseline (n=47,46,47,48,48,43,47) | 3.50 (1.32) | 3.96 (3.30) | 4.32 (2.74) | 4.65 (6.50) | 4.12 (2.44) | 3.90 (2.47) | 3.95 (2.30)
  Change at Week 1 (n=45,45,47,47,44,42,44) | 0.17 (1.63) | 0.60 (2.11) | 0.21 (2.50) | -0.27 (1.55) | -0.07 (1.26) | -0.51 (2.24) | -0.14 (2.00)
  Change at Week 2 (n=44,46,46,48,45,43,44) | 0.03 (1.40) | 1.04 (4.49) | 0.24 (3.08) | -0.44 (3.80) | -0.18 (1.01) | 0.04 (2.59) | 0.36 (2.96)
  Change at Week 4 (n=44,43,45,48,44,39,43) | 0.48 (2.14) | 0.61 (2.95) | -0.11 (2.31) | -0.30 (4.21) | 0.10 (1.50) | -0.08 (2.37) | 0.52 (2.43)
  Change at Week 6 (n=43,44,43,48,42,41,43) | 1.03 (4.65) | 0.36 (2.77) | -0.01 (2.46) | -0.71 (4.85) | 0.13 (1.45) | -0.21 (2.51) | 0.59 (3.32)
  Change at Week 8 (n=45,46,47,48,47,43,45) | 0.55 (2.19) | 0.51 (2.93) | -0.18 (2.30) | -0.04 (5.01) | 0.08 (1.50) | 0.31 (3.54) | 0.52 (3.07)

16. Secondary Outcome: Change From Baseline in Ocular Comfort Index (OCI) Score at Week 1, 2, 4, 6 and 8
Description: OCI: validated questionnaire to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contains 12 questions, each measured on a 7-point Likert scale ranging from 0 (never) to 6 (always/severe). Total score was transformed to range of 0 to 100, higher score indicated more ocular discomfort. Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 44 | 47
units on a scale
  Baseline (n=47,46,47,48,48,44,47) | 45.0 (7.66) | 43.9 (8.09) | 44.8 (7.69) | 46.0 (11.22) | 45.4 (8.41) | 42.3 (7.01) | 47.4 (12.51)
  Change at Week 1 (n=45,45,47,47,44,41,43) | -3.7 (7.28) | -5.9 (6.44) | -4.2 (6.49) | -3.9 (7.68) | -7.7 (9.99) | -4.3 (7.70) | -3.8 (7.79)
  Change at Week 2 (n=44,46,46,48,45,43,44) | -6.3 (7.89) | -6.0 (5.92) | -6.2 (9.00) | -5.9 (7.30) | -7.6 (9.89) | -4.4 (9.13) | -6.8 (10.59)
  Change at Week 4 (n=44,43,45,48,44,41,43) | -8.9 (8.44) | -7.6 (9.73) | -6.8 (8.58) | -5.7 (11.33) | -8.5 (10.88) | -6.1 (8.33) | -5.2 (8.23)
  Change at Week 6 (n=43,44,43,48,42,41,43) | -10.1 (9.75) | -9.1 (9.35) | -8.8 (7.46) | -7.5 (10.31) | -8.0 (9.72) | -7.3 (10.88) | -7.2 (9.36)
  Change at Week 8 (n=45,46,47,48,47,44,44) | -9.6 (8.98) | -9.9 (9.47) | -8.0 (8.81) | -7.4 (11.34) | -8.4 (9.42) | -8.8 (9.51) | -7.1 (10.16)

17. Secondary Outcome: Percentage of Participants With >= 5 Units Decrease in Total OCI Score
Description: OCI: validated questionnaire to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching. It contains 12 questions, each measured on a 7-point Likert scale ranging from 0 (never) to 6 (always/severe). Total score was transformed to range of 0 to 100, higher score indicated more ocular discomfort.
Time Frame: Week 1, 2, 4, 6, 8
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 46 | 47 | 48 | 47 | 44 | 44
percentage of participants
  Week 1 | 44.4 | 53.3 | 38.3 | 53.2 | 56.8 | 43.9 | 39.5
  Week 2 | 56.8 | 52.2 | 45.7 | 62.5 | 57.8 | 48.8 | 52.3
  Week 4 | 68.2 | 60.5 | 55.6 | 58.3 | 65.9 | 51.2 | 46.5
  Week 6 | 72.1 | 68.2 | 72.1 | 62.5 | 61.9 | 51.2 | 51.2
  Week 8 | 64.4 | 71.7 | 59.6 | 60.4 | 57.4 | 59.1 | 52.3

18. Secondary Outcome: Change From Baseline in Daily Artificial Tear Use at Week 1, 2, 4, 6 and 8
Description: Daily artificial tear use was assessed by collecting data on daily number of drops of artificial tear instilled in the eye using a participant diary. Decrease in daily artificial tear use indicated improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: drops/day
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 43 | 47
drops/day
  Baseline (n=47,46,47,48,48,43,47) | 3.4 (1.58) | 3.0 (1.63) | 3.0 (1.16) | 2.5 (1.65) | 3.0 (1.65) | 2.8 (1.20) | 2.9 (1.60)
  Change at Week 1 (n=45,46,47,48,47,43,45) | -0.7 (1.27) | -1.1 (0.99) | -0.8 (1.01) | -0.8 (1.01) | -0.9 (1.33) | -1.1 (1.01) | -0.6 (1.17)
  Change at Week 2 (n=44,46,45,48,47,42,44) | -0.9 (1.31) | -1.2 (1.09) | -0.8 (1.20) | -0.9 (0.99) | -0.9 (1.28) | -1.0 (1.03) | -0.6 (1.21)
  Change at Week 4 (n=44,44,45,48,45,41,44) | -1.1 (1.60) | -1.5 (1.22) | -0.9 (1.08) | -1.0 (0.95) | -0.9 (1.29) | -1.2 (1.27) | -0.8 (1.42)
  Change at Week 6 (n=44,44,46,48,43,40,43) | -1.5 (1.51) | -1.5 (1.08) | -0.9 (1.15) | -1.1 (1.07) | -1.0 (1.60) | -1.3 (1.10) | -0.7 (1.33)
  Change at Week 8 (n=46,46,47,48,47,43,46) | -1.2 (1.36) | -1.6 (1.20) | -1.0 (1.19) | -1.2 (1.04) | -1.1 (1.52) | -1.5 (1.27) | -0.9 (1.34)

19. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total and Subscale Score at Week 1, 2, 4, 6 and 8
Description: OSDI is a validated instrument for ocular surface disease. It has 12 items, each measured on 5-point Likert scale (0=none of the time, 4=all the time). Based on these item scores, a total OSDI score (question 1 [Q1]-Q12) and three subscale scores can be derived: Ocular Symptom (Q1-Q3), Vision-related function (Q4-Q9), and Environmental trigger (Q10-Q12). Each derived score ranges from 0 to 100, with a higher score indicates worse condition.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: ITT population. LOCF method was used for imputing missing data at Week 8. Here 'N' (number of participants analyzed) included those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 46 | 48 | 48 | 43 | 47
units on a scale
  Baseline:total (n=47,46,46,48,48,43,47) | 37.6 (21.46) | 35.6 (19.71) | 31.5 (17.95) | 41.8 (22.04) | 37.8 (18.76) | 35.6 (22.45) | 41.8 (22.93)
  Baseline:symptoms (n=47,46,46,48,48,43,47) | 39.7 (22.87) | 38.8 (21.60) | 38.6 (20.66) | 45.7 (24.37) | 41.7 (22.87) | 35.9 (20.86) | 47.3 (24.64)
  Baseline:function (n=46,46,45,48,47,43,44) | 31.8 (21.05) | 28.8 (20.30) | 23.5 (19.55) | 38.3 (26.66) | 31.8 (20.74) | 31.3 (27.07) | 36.1 (26.02)
  Baseline:triggers (n=46,41,42,45,42,41,43) | 46.7 (30.81) | 49.8 (29.64) | 42.0 (31.63) | 46.1 (29.64) | 45.6 (29.52) | 44.8 (26.92) | 50.3 (30.12)
  Change at Week 1:total (n=45,45,46,47,44,40,43) | -6.8 (14.39) | -5.1 (13.61) | -6.3 (13.79) | -8.9 (11.43) | -6.5 (17.18) | -9.2 (17.13) | -4.7 (12.46)
  Change at Week 1:symptoms (n=45,45,46,47,44,40,43) | -5.9 (16.73) | -4.1 (15.85) | -8.5 (17.52) | -8.2 (17.59) | -6.3 (20.26) | -6.9 (17.99) | -4.5 (13.03)
  Change at Week 1:function (n=43,45,44,47,43,39,39) | -6.1 (15.49) | -3.7 (16.32) | -4.4 (13.48) | -9.1 (14.77) | -4.4 (19.94) | -9.1 (17.81) | -7.3 (16.84)
  Change at Week 1:triggers (n=43,39,39,43,38,35,39) | -7.9 (23.64) | -12.0 (24.05) | -6.6 (24.74) | -10.2 (18.88) | -14.7 (23.12) | -15.0 (28.19) | -2.4 (18.97)
  Change at Week 2:total (n=44,46,45,48,45,43,44) | -8.7 (12.60) | -6.2 (12.09) | -8.6 (13.66) | -8.9 (13.08) | -4.7 (19.01) | -10.3 (20.16) | -7.3 (16.51)
  Change at Week 2:symptoms (n=44,46,45,48,45,43,44) | -9.1 (18.49) | -6.2 (13.99) | -11.5 (17.79) | -11.5 (18.12) | -6.9 (19.41) | -9.7 (21.74) | -7.6 (17.77)
  Change at Week 2:function (n=42,46,42,48,43,43,41) | -8.6 (14.26) | -5.8 (13.67) | -5.5 (12.92) | -7.6 (16.52) | -3.5 (23.92) | -7.0 (19.10) | -8.6 (19.44)
  Change at Week 2:triggers (n=42,40,40,38,35,39,40) | -9.9 (18.38) | -7.9 (24.98) | -8.8 (24.76) | -9.4 (16.60) | -10.1 (29.00) | -19.2 (29.05) | -5.5 (21.42)
  Change at Week 4:total (n=44,43,44,48,44,41,43) | -11.5 (15.88) | -7.2 (12.98) | -8.1 (15.53) | -9.7 (14.12) | -10.0 (20.92) | -11.3 (17.12) | -7.0 (13.95)
  Change at Week 4:symptoms (n=44,43,44,48,44,41,43) | -12.1 (18.19) | -8.5 (12.79) | -13.4 (20.27) | -10.9 (18.37) | -10.8 (23.47) | -10.4 (18.61) | -6.6 (15.06)
  Change at Week 4:function (n=43,42,42,47,41,41,40) | -10.2 (16.42) | -4.7 (15.98) | -6.3 (16.97) | -8.5 (16.77) | -5.1 (20.37) | -7.3 (18.75) | -8.7 (17.83)
  Change at Week 4:triggers (n=43,36,39,43,36,37,39) | -13.5 (26.02) | -10.4 (21.90) | -5.8 (30.16) | -9.8 (23.23) | -16.3 (29.55) | -21.5 (25.07) | -4.7 (20.90)
  Change at Week 6:total (n=43,44,42,48,42,41,43) | -10.5 (14.26) | -9.1 (14.19) | -7.9 (13.89) | -10.9 (14.33) | -8.1 (20.48) | -14.0 (19.43) | -7.7 (14.00)
  Change at Week 6:symptoms (n=43,44,42,48,42,41,43) | -11.2 (18.36) | -10.0 (13.76) | -12.3 (17.96) | -11.4 (19.52) | -7.1 (21.03) | -13.4 (21.80) | -9.1 (15.52)
  Change at Week 6:function (n=42,44,38,46,40,41,40) | -9.1 (18.88) | -7.0 (15.30) | -5.1 (14.46) | -9.6 (14.74) | -3.7 (20.10) | -9.3 (19.34) | -8.3 (17.09)
  Change at Week 6:triggers (n=40,38,37,41,34,38,39) | -13.2 (21.62) | -13.0 (24.80) | -9.7 (23.61) | -9.2 (24.85) | -12.4 (32.88) | -24.5 (28.3) | -5.9 (22.65)
  Change at Week 8:total (n=45,46,46,48,32,35,39) | -11.0 (18.55) | -8.5 (15.34) | -7.6 (15.22) | -8.8 (16.56) | -9.5 (20.92) | -12.7 (18.21) | -6.6 (16.11)
  Change at Week 8:symptoms (n=45,46,46,48,47,43,44) | -13.1 (20.37) | -8.9 (16.14) | -11.6 (20.52) | -11.6 (20.68) | -10.5 (23.98) | -14.3 (21.54) | -7.4 (17.72)
  Change at Week 8:function (n=44,46,45,48,46,43,41) | -9.1 (21.31) | -6.4 (16.54) | -4.5 (14.82) | -9.2 (18.33) | -6.2 (23.86) | -9.2 (18.31) | -6.8 (19.72)
  Change at Week 8:triggers(n=44,41,42,45,,41,41,41) | -12.2 (24.86) | -14.2 (24.46) | -8.4 (23.62) | -6.4 (29.08) | -13.5 (29.07) | -19.6 (26.06) | -4.8 (23.62)

20. Secondary Outcome: Percentage of Participants With >= 10 Units Decrease in Total OSDI Score
Description: OSDI is a validated instrument for ocular surface disease. It has 12 items, each has a raw score measured on 5-point Likert scale (0=none of the time, 4=all the time). Based on these item scores, a total OSDI score can be derived which ranges from 0 to 100; a higher score indicates worse ocular disease.
Time Frame: Week 1, 2, 4, 6, 8
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 45 | 46 | 46 | 48 | 47 | 43 | 44
percentage of participants
  Week 1 | 37.8 | 37.8 | 34.8 | 46.8 | 45.5 | 40.0 | 37.2
  Week 2 | 50.0 | 45.7 | 40.0 | 43.8 | 33.3 | 39.5 | 43.2
  Week 4 | 47.7 | 44.2 | 38.6 | 50.0 | 45.5 | 41.5 | 44.2
  Week 6 | 46.5 | 52.3 | 35.7 | 52.1 | 40.5 | 51.2 | 39.5
  Week 8 | 40.0 | 50.0 | 41.3 | 47.9 | 44.7 | 46.5 | 38.6

21. Secondary Outcome: Change From Baseline Ocular Surface Disease Index (OSDI) Raw Score at Week 1, 2, 4, 6 and 8
Description: OSDI is a validated instrument for ocular surface disease. It has 12 items, each with a raw score measured on 5-point Likert scale (0=none of the time, 4=all the time).
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: Data for OSDI raw score was not analyzed due to the exploratory nature and overwhelming amount of data derived from the analysis.
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Modified Ocular Comfort Index (mOCI) Raw Scores at Week 1, 2, 4, 6 and 8
Description: mOCI consisted of the original 12-item OCI plus additional questions on other dry eye symptoms and their impact to participant's life. Each item was measured on a 7-point Likert scale ranging from 0 (never) to 6 (always/severe). Negative change from baseline indicated improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, 8
Population: Data for mOCI raw score was not analyzed due to the exploratory nature and overwhelming amount of data derived from the analysis.
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in National Eye Institute Visual Functioning Questionnaire 25-item Score (NEI-VFQ-25) at Week 8
Description: NEI-VFQ-25 questionnaire included 25 items based on which overall composite VFQ score and 12 subscales were derived: general health (GH), general vision (GV), ocular pain (OP), near activities (NAct), distance activities (DA), social functioning (SF), mental health (MH), role difficulties (RD), dependency, driving, color vision (CV) and peripheral vision (PV). Response to each question converted to 0-100 score. Each subscale, total score=average of items contributing to score. For each subscale and total score, score range: 0 to 100, higher score=less symptoms/better visual functioning.
Time Frame: Baseline, Week 8
Population: ITT population included all enrolled participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Number analyzed (Participants) | 47 | 46 | 47 | 48 | 48 | 43 | 47
Units on a scale
  Baseline: GH (n=46,46,47,48,48,43,47) | 65.22 (20.74) | 66.85 (21.12) | 62.77 (20.10) | 66.15 (24.99) | 59.90 (23.49) | 66.86 (25.43) | 57.98 (20.92)
  Baseline: GV (n=47,46,47,48,48,43,47) | 72.77 (16.38) | 75.65 (12.59) | 73.62 (14.51) | 72.50 (20.05) | 72.08 (13.52) | 70.70 (17.10) | 73.19 (13.37)
  Baseline: OP (n=47,46,47,48,48,43,47) | 59.31 (18.70) | 59.51 (18.85) | 61.17 (20.89) | 53.65 (23.06) | 55.47 (19.28) | 56.40 (17.76) | 50.27 (24.76)
  Baseline: NAct (n=47,46,47,48,48,43,47) | 68.62 (18.49) | 70.92 (17.53) | 76.60 (18.60) | 64.41 (23.36) | 66.06 (20.01) | 72.00 (21.53) | 64.36 (23.36)
  Baseline: DA (n=47,46,47,48,48,43,47) | 73.76 (17.63) | 77.36 (17.71) | 81.38 (16.32) | 72.05 (25.12) | 73.00 (17.13) | 71.90 (20.66) | 69.33 (21.92)
  Baseline: SF (n=47,46,47,48,48,43,47) | 89.10 (14.89) | 93.21 (10.77) | 93.88 (11.62) | 86.46 (21.39) | 89.84 (14.51) | 87.79 (18.99) | 85.64 (20.52)
  Baseline: MH (n=47,46,47,48,48,43,47) | 72.34 (24.55) | 73.23 (19.88) | 77.53 (19.71) | 64.84 (26.13) | 67.97 (22.94) | 72.67 (22.24) | 70.35 (23.73)
  Baseline: RD (n=47,46,47,48,48,43,47) | 68.09 (23.28) | 72.83 (20.12) | 76.33 (25.96) | 61.98 (29.73) | 67.71 (26.02) | 68.02 (26.91) | 68.09 (27.81)
  Baseline:dependency (n=47,45,47,47,48,43,47) | 88.48 (21.46) | 93.89 (10.42) | 94.33 (11.54) | 81.91 (25.79) | 88.02 (23.34) | 87.79 (22.15) | 89.72 (19.90)
  Baseline:driving (n=46,44,45,46,41,41,44) | 73.64 (17.15) | 76.89 (15.65) | 77.22 (19.09) | 78.44 (20.38) | 71.54 (22.28) | 71.65 (21.23) | 71.12 (19.80)
  Baseline: CV (n=46,46,47,48,48,43,47) | 89.67 (21.46) | 96.20 (9.08) | 93.62 (13.26) | 90.10 (18.41) | 93.75 (14.12) | 91.28 (17.15) | 90.43 (17.72)
  Baseline: PV (n=47,46,46,48,46,43,47) | 77.13 (23.21) | 82.61 (20.32) | 85.87 (21.51) | 80.21 (25.24) | 79.89 (21.49) | 79.65 (26.31) | 80.32 (22.68)
  Baseline: Overall (n=47,46,47,48,48,43,47) | 75.62 (14.43) | 79.30 (10.95) | 81.08 (12.99) | 73.19 (19.31) | 75.06 (13.96) | 75.40 (15.58) | 73.97 (16.76)
  Change at Week 8: GH (n=42,43,44,48,41,40,41) | 0.00 (13.53) | -2.91 (14.65) | 0.00 (15.25) | 2.08 (19.18) | 1.22 (18.50) | -0.63 (14.42) | 1.83 (10.29)
  Change at Week 8: GV (n=43,43,44,48,41,40,41) | 1.86 (16.22) | 1.86 (12.20) | 1.36 (7.95) | 3.75 (12.82) | 1.46 (18.11) | 5.00 (15.53) | -0.49 (10.48)
  Change at Week 8: OP (n=43,43,44,48,41,40,41) | 15.12 (19.59) | 11.63 (21.89) | 13.35 (20.95) | 9.38 (15.79) | 11.59 (19.24) | 16.56 (20.88) | 9.45 (19.72)
  Change at Week 8: NAct (n=43,43,44,48,41,40,41) | 7.17 (17.21) | 8.62 (15.33) | 4.17 (12.64) | 7.12 (16.49) | 10.87 (19.07) | 7.40 (15.49) | 9.96 (19.65)
  Change at Week 8: DA (n=43,43,44,48,41,40,41) | 6.78 (12.50) | 5.43 (13.22) | 3.03 (13.46) | 4.43 (11.32) | 8.84 (17.88) | 8.85 (17.66) | 5.89 (14.67)
  Change at Week 8: SF (n=43,43,44,48,41,40,41) | 3.20 (12.82) | 2.62 (11.75) | 2.27 (10.54) | 3.39 (13.58) | 5.79 (13.43) | 6.88 (18.55) | 8.23 (12.06)
  Change at Week 8: MH (n=43,43,44,48,41,40,41) | 10.61 (19.27) | 9.59 (17.27) | 4.55 (13.57) | 5.34 (15.95) | 11.28 (18.92) | 10.63 (22.30) | 5.95 (16.41)
  Change at Week 8: RD (n=43,43,44,48,41,40,41) | 6.98 (15.74) | 5.52 (27.59) | 4.55 (20.37) | 5.47 (18.93) | 8.23 (24.94) | 12.50 (25.94) | 0.00 (29.05)
  Change Week 8:dependency(n=43,42,44,47,41,40,41) | 7.56 (21.32) | 1.19 (15.79) | 1.89 (8.96) | 4.61 (14.83) | 5.39 (19.59) | 7.08 (17.45) | 2.24 (11.94)
  Change at Week 8:driving (n=42,41,42,46,33,38,39) | 6.15 (14.47) | 3.46 (16.24) | 3.27 (13.64) | 0.36 (12.29) | 3.91 (14.43) | 8.22 (13.65) | 3.95 (13.07)
  Change at Week 8: CV (n=42,43,44,48,41,40,41) | 4.76 (13.79) | 2.33 (9.15) | 3.98 (10.71) | 2.08 (16.97) | 2.44 (13.47) | 5.63 (19.19) | 4.88 (16.03)
  Change at Week 8: PV (n=43,43,44,48,39,40,41) | 11.05 (22.03) | 4.07 (15.36) | 1.70 (15.62) | 3.65 (18.59) | 6.41 (21.24) | 6.88 (20.40) | 6.71 (20.17)
  Change at Week 8: Overall (n=43,43,44,48,41,40,41) | 7.44 (9.55) | 5.13 (9.20) | 3.98 (7.44) | 4.50 (8.19) | 7.15 (11.60) | 8.67 (11.50) | 5.15 (10.42)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo Twice Daily | CP-690,550, 0.0003% Twice Daily | CP-690,550, 0.001% Twice Daily | CP-690,550, 0.003% Twice Daily | CP-690,550, 0.005% Twice Daily | CP-690,550, 0.005% Once Daily | Restasis Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/46 | 0/47 | 1/48 | 1/48 | 1/44 | 1/47
Other Adverse Events (participants affected / at risk) | 23/47 | 11/46 | 22/47 | 21/48 | 15/48 | 15/44 | 26/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Twice Daily (N=47) | CP-690,550, 0.0003% Twice Daily (N=46) | CP-690,550, 0.001% Twice Daily (N=47) | CP-690,550, 0.003% Twice Daily (N=48) | CP-690,550, 0.005% Twice Daily (N=48) | CP-690,550, 0.005% Once Daily (N=44) | Restasis Twice Daily (N=47)
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Twice Daily (N=47) | CP-690,550, 0.0003% Twice Daily (N=46) | CP-690,550, 0.001% Twice Daily (N=47) | CP-690,550, 0.003% Twice Daily (N=48) | CP-690,550, 0.005% Twice Daily (N=48) | CP-690,550, 0.005% Once Daily (N=44) | Restasis Twice Daily (N=47)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye, BOTH EYES (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Asthenopia, BOTH EYES (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Blepharitis, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract nuclear, BOTH EYES (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival cyst, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia, BOTH EYES (Eye disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1
Conjunctival hyperaemia, FELLOW EYE ONLY (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Conjunctival hyperaemia, STUDY EYE ONLY (Eye disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0
Conjunctival oedema, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival oedema, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival oedema, STUDY EYE ONLY (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Corneal deposits, BOTH EYES (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corneal disorder, BOTH EYES (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corneal disorder, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal epithelium defect, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal erosion, BOTH EYES (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Corneal oedema, STUDY EYE ONLY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye, BOTH EYES (Eye disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Erythema of eyelid, STUDY EYE ONLY (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Excessive eye blinking, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye disorder, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation, BOTH EYES (Eye disorders) | 1 | 1 | 1 | 2 | 2 | 0 | 1
Eye irritation, FELLOW EYE ONLY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain, BOTH EYES (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 1
Eye pain, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus, BOTH EYES (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Eye pruritus, FELLOW EYE ONLY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling, BOTH EYES (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eyelid disorder, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid irritation, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid irritation, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid margin crusting, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid oedema, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foreign body sensation in eyes, BOTH EYES (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Iritis, BOTH EYES (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased, BOTH EYES (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Lacrimation increased, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Meibomian gland dysfunction, BOTH EYES (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Meibomian gland dysfunction, FELLOW EYE ONLY (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Meibomian gland dysfunction, STUDY EYE ONLY (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2
Myodesopsia, FELLOW EYE ONLY (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myodesopsia, STUDY EYE ONLY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ocular hyperaemia, BOTH EYES (Eye disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 1
Ocular hyperaemia, STUDY EYE ONLY (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Punctate keratitis, BOTH EYES (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Punctate keratitis, STUDY EYE ONLY (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Trichiasis, FELLOW EYE ONLY (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred, BOTH EYES (Eye disorders) | 1 | 0 | 1 | 2 | 2 | 1 | 1
Visual acuity reduced, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced, FELLOW EYE ONLY (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced, STUDY EYE ONLY (Eye disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment, BOTH EYES (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Instillation site pain, BOTH EYES (General disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 3
Instillation site pain, STUDY EYE ONLY (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Instillation site pruritus, BOTH EYES (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sensation of foreign body, FELLOW EYE ONLY (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Temperature intolerance, BOTH EYES (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity, BOTH EYES (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis bacterial, STUDY EYE ONLY (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perichondritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contact lens complication, BOTH EYES (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal abrasion, STUDY EYE ONLY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foreign body trauma, FELLOW EYE ONLY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superficial injury of eye, STUDY EYE ONLY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation, BOTH EYES (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Telangiectasia, STUDY EYE ONLY (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired work ability, BOTH EYES (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection, BOTH EYES (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In this study, a variance was made in the planned analysis. At the time of data analysis, results from Stage 1 and 2 were combined for efficacy and safety analyses. Hence, results are presented together for both stages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.